CLINICAL TRIAL: NCT04267744
Title: Usability and Utility Assessment of Passive Remote Monitoring of Multiple Novel Indicators of Heart Failure
Brief Title: Remote Monitoring of Multiple Indicators of Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Washington University School of Medicine (Other)
Collaborators: Healthcare Innovation Lab (Unknown); MYIA Labs, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201908180
Record Dates: First submitted 2020-02-05; First posted 2020-02-13 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure
Keywords: NYHA II-IV; Reduced Ejection Fraction; Cardiology
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Device: Myia Health platform and in-home suite of devices®
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote patient monitoring (Other): After consenting to the study, the Myia in-home suite of devices, and mobile phone application if the patient owns a smart phone, will be provided to all recruited patients. The data flowing from the Myia platform will be available to clinicians and patients for the duration of the pilot and utilized to complete study activities.
  Patients enrolled will transmit daily vital sign data to the Myia Health remote patient monitoring platforms for clinical review.
  Enrolled patients will complete medication change/compliance survey monthly to assess for medication changes.
  Enrolled patients will complete symptomatic assessments (KCCQ-12) at 0, 3, and 6 months.
  Enrolled patients will complete a Check-In survey to assess utility and usability of the intervention at the 2, 4, and 6 month timepoints
  Interventions: Other: Myia Health® remote patient monitoring unblinded treatment arm

INTERVENTIONS:
Other: Myia Health® remote patient monitoring unblinded treatment arm — After consenting to the study, the Myia in-home suite of devices will be provided to all recruited patients. The data flowing from the Myia platform will be available to clinicians and patients for the duration of the pilot and utilized to complete study activities.
  Device: Myia Health platform and in-home suite of devices®:
  Emfit Ballistocardiograph® Withings Connected Scale® VitalScout (VivaLink) ECG Accelerometer® Omron Blood Pressure Monitor® (Sphygmomanometer) Cradlepoint - Hotspot / Adaptor® (LTE Connection) Samsung Galaxy Tab A 8.0"® (User Interface)
  Other Names: Myia Health platform and in-home suite of devices®

SUMMARY:
This study is intended to evaluate the impact of passive continuous remote patient monitoring to assist in the outpatient management of heart failure (HF) patients.

DETAILED DESCRIPTION:
The study will prospectively evaluate the usability, utility, and efficacy of remote monitoring using novel noninvasive technologies in HF patients in an outpatient setting. Investigators will gather dynamic, longitudinal data from multiple sensors, in addition to patient-reported and physician-reported data. Both the patient interface through interactions with the sensors and mobile application, and the clinician interface through the monitoring portal, will be evaluated for usability, utility and efficacy.

Patients will be recruited for the study from the Barnes Jewish Hospital Advanced Heart Failure Clinic. Eligible individuals will receive onboarding instructions and a study schedule detailing the required surveys and clinical activities they will be asked to complete over a period of 7 months. In addition to onboarding instructions and a study schedule, individuals will have the kit of sensors shipped to their home.

After the Myia Home Hub and Myia Sensor Suite are set up, data will begin to be transmitted. Following a run in period where data is collected and delivered but not acted upon by clinicians all eligible participants will move forward with 6 month interactive study monitoring.

In addition to obtaining questionnaires and using the devices in the Myia kit, participants will also be asked to obtain their blood pressure and weight daily.

During the course of the study, outpatient health status data for the group will be collected, summarized and delivered to clinicians in an electronic dashboard. The format and content of the data dashboard will be updated based on user feedback throughout the study. Required changes deemed appropriate by the healthcare team will be incorporated into the software platform alongside any standard updates.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients cared for by BJH Advanced Heart Failure Clinic, where BJH is their primary cardiology care team
2. Age ≥ 18 years old at time of consent
3. HFrEF diagnosis in the BJH Advanced Heart Failure Clinic medical record
4. Has had an ER presentation or hospitalization related to their heart failure in last 12 months prior to enrollment
5. Most recent recorded Left Ventricular Ejection Fraction (LVEF) of < 50% and at least 1 recorded LVEF of < 40%
6. Scheduled clinic visit 90- 180 days after study enrollment.
7. NYHA Class II-IV
8. Sleeps in the same bed at ≥ 4 days per week
9. Able to ambulate
10. Willingness to complete the required surveys, measurements and study activities

Exclusion Criteria:

1. Current ventricular assist device or cardiac transplant.
2. Currently listed for cardiac transplantation
3. End-Stage Renal Disease on chronic dialysis
4. Malignancy diagnosis undergoing active treatment
5. Hospice or palliative care
6. Living in a skilled nursing facility or other chronic care facility (ambulatory patients only)
7. Self-reported pregnancy or planned pregnancy in the next 6 months
8. Inability or unwillingness to consent and/or follow requirements of the study
9. Planned major surgeries or procedures requiring hospitalization in next 6 months
10. Use of Lifevest or other worn device that may affect ballistocardiogram measurements
11. Patient weight > 385 lbs at time of enrollment
12. Life expectancy <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Myia Platform feasibility: questionnaire | From baseline to 6 months (final)
  Patient perception of the Myia Platform will be assessed during the study using a structured questionnaire, delivered either electronically or by paper to patients by research staff.
  Patient Platform satisfaction/usability/utility questionnaire: The formal title of the questionnaire is 'Check In Survey' and it consists of 17 questions with scaled options, 1-7 (1=most positive, 7=most negative) and it is administered at 3 time points. The lower the overall total the more positive the patient rating of the Myia Platform.

SECONDARY OUTCOMES:
Persistence of minimally useful data acquisition of a remote patient monitoring platform to monitor the health status of patients living with heart failure. | From baseline to 6 months time (final)
  Acquisition of minimally useful data profile: Weeks where minimally useful data profile collected/total number of weeks. This endpoint will be defined retrospectively by the clinical team.
Persistence of daily data acquisition of a remote patient monitoring platform to monitor the health status of patients living with heart failure. | From baseline to 6 months time (final)
  Acquisition of any data point daily: Days with >1 data point collected/total number of days
Persistence of weekly data acquisition of a remote patient monitoring platform to monitor the health status of patients living with heart failure. | From baseline to 6 months time (final)
  Acquisition of any data point weekly: Weeks with >1 data point collected/total number of weeks
Persistence of vital sign data acquisition of a remote patient monitoring platform to monitor the health status of patients living with heart failure. | From baseline to 6 months time (final)
  Acquisition of continuous vital sign data variables daily: Days with >1 data point collected/total number of days
Persistence of greater than 1 data point per week data acquisition of a remote patient monitoring platform to monitor the health status of patients living with heart failure. | From baseline to 6 months time (final)
  Acquisition of continuous data variables weekly: Weeks with >1 data point collected/total number of weeks
Medication management: total number of medication changes | From baseline to 6 months time (final)
  Absolute count of heart failure medication changes per patient. This metric will be calculated on a per patient level. Any change in dose or frequency of medication will be considered a medication change.
Medication management: length of time to medication change | From baseline to 6 months time (final)
  Mean time to heart failure medication change per patient. Average time interval between a change to 1 or more heart failure drugs between the baseline and 6 month time points.
Medication management: target dose | From baseline to 6 months time (final)
  Distance from target dose of heart failure medication (< 50% target dose, 50%-75% of target dose, 75%-100% of target dose)
  The baseline use and dose of the following heart failure medication categories will be examined for each patient at baseline:
  Beta Blockers Digoxin ACE, ARB, ARNIs Hydralazine Nitrates Loop Diuretics Aldosterone Antagonists For each medication class, the presence and absence of absolute contraindications will be determined based on documentation in the medical record or as ascertained by study investigators. For each patient and each medication, available dose information will be reviewed in reference to recommended target doses by clinical practice guidelines. Distance to target dose will be assessed at baseline and follow-up. The difference in the relative proportion of people in the target dose categories will be compared between treatment and usual care groups.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Ewald, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Background] Chen J, Normand SL, Wang Y, Krumholz HM. National and regional trends in heart failure hospitalization and mortality rates for Medicare beneficiaries, 1998-2008. JAMA. 2011 Oct 19;306(15):1669-78. doi: 10.1001/jama.2011.1474. PMID 22009099
- [Background] Wolfel EE. Can we predict and prevent the onset of acute decompensated heart failure? Circulation. 2007 Oct 2;116(14):1526-9. doi: 10.1161/CIRCULATIONAHA.107.729608. No abstract available. PMID 17909113
- [Background] Ping W, Jin-Gang W, Xiao-Bo S, Wei H. The research of telemedicine system based on embedded computer. Conf Proc IEEE Eng Med Biol Soc. 2005;2006:114-7. doi: 10.1109/IEMBS.2005.1616355. PMID 17282124
- [Background] Abraham WT, Adamson PB, Bourge RC, Aaron MF, Costanzo MR, Stevenson LW, Strickland W, Neelagaru S, Raval N, Krueger S, Weiner S, Shavelle D, Jeffries B, Yadav JS; CHAMPION Trial Study Group. Wireless pulmonary artery haemodynamic monitoring in chronic heart failure: a randomised controlled trial. Lancet. 2011 Feb 19;377(9766):658-66. doi: 10.1016/S0140-6736(11)60101-3. PMID 21315441
- [Background] Boehmer JP, Hariharan R, Devecchi FG, Smith AL, Molon G, Capucci A, An Q, Averina V, Stolen CM, Thakur PH, Thompson JA, Wariar R, Zhang Y, Singh JP. A Multisensor Algorithm Predicts Heart Failure Events in Patients With Implanted Devices: Results From the MultiSENSE Study. JACC Heart Fail. 2017 Mar;5(3):216-225. doi: 10.1016/j.jchf.2016.12.011. PMID 28254128
- [Background] Weng SF, Reps J, Kai J, Garibaldi JM, Qureshi N. Can machine-learning improve cardiovascular risk prediction using routine clinical data? PLoS One. 2017 Apr 4;12(4):e0174944. doi: 10.1371/journal.pone.0174944. eCollection 2017. PMID 28376093
- [Background] Chan PS, Oetgen WJ, Spertus JA. The Improving Continuous Cardiac Care (IC(3)) program and outpatient quality improvement. Am J Med. 2010 Mar;123(3):217-9. doi: 10.1016/j.amjmed.2009.09.019. No abstract available. PMID 20193826
- [Background] Ong MK, Romano PS, Edgington S, Aronow HU, Auerbach AD, Black JT, De Marco T, Escarce JJ, Evangelista LS, Hanna B, Ganiats TG, Greenberg BH, Greenfield S, Kaplan SH, Kimchi A, Liu H, Lombardo D, Mangione CM, Sadeghi B, Sadeghi B, Sarrafzadeh M, Tong K, Fonarow GC; Better Effectiveness After Transition-Heart Failure (BEAT-HF) Research Group. Effectiveness of Remote Patient Monitoring After Discharge of Hospitalized Patients With Heart Failure: The Better Effectiveness After Transition -- Heart Failure (BEAT-HF) Randomized Clinical Trial. JAMA Intern Med. 2016 Mar;176(3):310-8. doi: 10.1001/jamainternmed.2015.7712. PMID 26857383
- [Background] Krumholz HM, Merrill AR, Schone EM, Schreiner GC, Chen J, Bradley EH, Wang Y, Wang Y, Lin Z, Straube BM, Rapp MT, Normand SL, Drye EE. Patterns of hospital performance in acute myocardial infarction and heart failure 30-day mortality and readmission. Circ Cardiovasc Qual Outcomes. 2009 Sep;2(5):407-13. doi: 10.1161/CIRCOUTCOMES.109.883256. Epub 2009 Jul 9. PMID 20031870
- [Background] Chun S, Tu JV, Wijeysundera HC, Austin PC, Wang X, Levy D, Lee DS. Lifetime analysis of hospitalizations and survival of patients newly admitted with heart failure. Circ Heart Fail. 2012 Jul 1;5(4):414-21. doi: 10.1161/CIRCHEARTFAILURE.111.964791. Epub 2012 May 2. PMID 22556322
- [Background] Tung YC, Chou SH, Liu KL, Hsieh IC, Wu LS, Lin CP, Wen MS, Chu PH. Worse Prognosis in Heart Failure Patients with 30-Day Readmission. Acta Cardiol Sin. 2016 Nov;32(6):698-707. doi: 10.6515/acs20151113a. PMID 27899857
- [Background] Sud M, Yu B, Wijeysundera HC, Austin PC, Ko DT, Braga J, Cram P, Spertus JA, Domanski M, Lee DS. Associations Between Short or Long Length of Stay and 30-Day Readmission and Mortality in Hospitalized Patients With Heart Failure. JACC Heart Fail. 2017 Aug;5(8):578-588. doi: 10.1016/j.jchf.2017.03.012. Epub 2017 May 10. PMID 28501521
- [Background] Holland R, Rechel B, Stepien K, Harvey I, Brooksby I. Patients' self-assessed functional status in heart failure by New York Heart Association class: a prognostic predictor of hospitalizations, quality of life and death. J Card Fail. 2010 Feb;16(2):150-6. doi: 10.1016/j.cardfail.2009.08.010. Epub 2009 Oct 22. PMID 20142027
- [Background] Soto GE, Jones P, Weintraub WS, Krumholz HM, Spertus JA. Prognostic value of health status in patients with heart failure after acute myocardial infarction. Circulation. 2004 Aug 3;110(5):546-51. doi: 10.1161/01.CIR.0000136991.85540.A9. Epub 2004 Jul 19. PMID 15262843
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] Greene SJ, Fonarow GC, Butler J. Reply: Titration of Guideline-Directed Medical Therapy Improves Patient-Centered Outcomes in Heart Failure With Reduced Ejection Fraction. J Am Coll Cardiol. 2019 Sep 10;74(10):1426-1427. doi: 10.1016/j.jacc.2019.06.061. No abstract available. PMID 31488284